#### CONFIDENTIAL AND PROPRIETARY

Information provided herein is the property of the University-Hospital of Brescia. Nothing herein is to be reproduced, published, or disclosed to others in any way without the prior expressed written permission of the University-Hospital of Brescia.

Title of Study: Efficacy of guided biofilm therapy in paediatric patient: a randomized clinical trial

Type of Study: Clinical

Protocol No: PROTOCOL # BABYPLAK NP 5675

Sponsor: ASST Spedali Civili di Brescia

Expected study start date: GEN, 2023 (study initiation)

Study Location/Country: Brescia, Italy

# **Test Products w/ PDM Numbers:**

CE marked Medical Device to be used as an adjunct therapy to standard in pediatric patients (Confidential information).

Study Title: Efficacy of guided biofilm therapy (GBT) in paediatric patient: a

randomized clinical trial.

Study sites:

ASST Spedali Civili di Brescia

University of Brescia

Brescia, Italy.

Study Phase: IV.

Name of Medical Device: Plus Powder® and Biofilm Discloser® (EMS Electrical Medical

Systems SA, CH 1260-Nyon, Switzerland)

Objective: The objective of the clinical study is to assess the efficacy of

disclosing plaque agent and erythritol powder to remove biofilm and

plaque in pediatric patient during professional oral hygiene.

Patient Population: 120 pediatric subject, systemically healthy (ASA I e II), male and

female (6 – 12 years), with at least 80% of dental formula and with

at least 8/12 frontal dental elements.

Structure: Parallel arms: Number of treatments: 4

- Guided biofilm therapy with disclosing plaque (GBT+)

- Guided biofilm therapy without disclosing plaque (GBT-)

- Ultrasonic debridement with disclosing plaque (US+C+)

- Ultrasonic debridement without disclosing plaque (US+C-)

Duration of study: 36 months.

36 months enrolment

Number of Centers: One.

Method of Patient Selection: pediatric patients who require professional oral hygiene

Total Sample Size: 120 pediatric subjects will be recruited (randomized) to participate

in this study, with 120 expected to complete the study.

Primary Efficacy Variable: Primary outcome measure will be the percentage of area in which

the disclosing plaque agent is present (RPA: Residual Plaque

Area) in all groups after professional oral hygiene

# Efficacy of guided biofilm therapy (GBT) in pediatric patient: a randomized clinical trial. PROTOCOL #BABYPLAK

Protocol Date: OCT 10, 2022

# **Protocol Approval**

Signature Page

\_\_\_\_\_

Date

# Responsibilities

The **principal investigator's** responsibilities are described in detail in ISO norm 14155:2011 for the clinical investigation of medical devices for human subjects.

The role of the principal investigator is to implement and manage the day-to-day conduct of the clinical investigation as well as ensure data integrity and the rights, safety and well-being of the subjects involved in the clinical investigation.

The principal investigator shall be qualified by education, training and experience to assume responsibilities for the proper conduct of the clinical investigation. In particular, the principal investigator is responsible for:

- qualification of investigation site;
- communication with Ethics Committee;
- compliance with Informed Consent process;
- compliance with Clinical Investigation Plan.

Under the direct supervision of the Principal Investigator, certain duties may be delegated during the course of the study. These responsibilities will be documented on the transfer of responsibilities form maintained in the Investigator Site file.

The **Statistician** will be responsible for:

- sample size calculation;
- statistical plan;
- statistical section of the protocol;
- statistical evaluation;
- final statistical report.

#### **OBJECTIVE**

The study will be performed to assess the efficacy of disclosing plaque agent (DPA) and erythritol powder to remove biofilm and plaque in pediatric patient during professional oral hygiene.

#### INTRODUCTION

In the mouth of the patients the biofilm is not always evident, so it's removal can be difficult.

Using the disclosing plaque agent before the therapy as a guide to remove the biofilm may be a solution. Thanks to this tool, we can clearly see where the plaque is, so it's removal can be easier. In pediatric patients is more difficult to remove biofilm and plaque cause of less collaboration to a correct oral hygiene. Probably, using a disclosing plaque agent that guide the operator, could give more security and faster for a better removal of the biofilm. Moreover, the use of low abrasiveness powder could lead to several advantages like a decrease of patients' uncomfortable feeling, the shortest execution time and the possibility of cleaning areas with difficult access and the less damage on soft and hard tissue respect the traditional professional oral hygiene.

For this reasons, we decided to study the efficacy of this method.

#### STUDY OUTCOMES

Primary outcome measure: comparison between groups of the percentage of area in which the disclosing plaque agent is present (RPA: Residual Plaque Area).

RPA: residual plaque area: percentage of area with residual plaque coloured by disclosing plaque agent. This will be calculated with a ImageJ Software.

Secondary outcome measure:

- comparison between groups of FMPS (Full Mouth Plaque Score) after professional oral hygiene – clinical parameter
- comparison between groups on execution time
- · comparison between groups about feeling of patient ad operator

#### STUDY POPULATION

One hundred and twenty (120) children, aged 6-12 years, will be entered into study (randomized). It is expected that forty (120) subjects will complete the study.

Randomized subjects who deviate from the protocol (major protocol deviation) and, for this reason, are excluded from the analysis, will be replaced to guarantee that the sample required for the analysis (120) is reached.

Patient will be treated at the Department of Surgical Specialities Radiological Science and Public Health, School of Dentistry, Section of Periodontics, Brescia, Italy from 01/2023.

# **Inclusion Characteristics**

- Signed Informed Consent Form (pediatric patient and parent).
- Male and female subjects, aged 6 -12 years, inclusive.
- Good general health (ASA I e II)
- With at least 80% of dental formula
- With at least 8/12 frontal dental elements.

#### **Exclusion Characteristics**

- Not willing to follow the agreed protocol.
- Presence of orthodontic appliances.
- Tumors or significant pathology of the soft or hard tissues of the oral cavity.
- Current radiotherapy or chemotherapy.
- History of allergy to Erythritol.
- History of adverse reactions to lactose or fermented milk products.

A written informed consent will be obtained from each included patient after explanation of the risks and benefits of participating to this study. No change in the trial design will be made after approval of the Ethical Committee.

#### 1. STUDY DESIGN

The study design was chosen according to the current standards required by GCP and according to national requirements.

- a. A 2 by 2 parallel design.
- b. The RCT will be run as mono-center;
- c. A total of 120 subjects will be recruited to participate in the study. It is expected that all of 120 subjects will complete the study in total;
- d. Admission into the study will be via rolling admission (estimated recruitment time: 36 months);
- e. Each subject must be pediatric patient who needs a professional oral hygiene;
- a. Each subject will follow the following treatment protocol:
  - i. Visit (T0): consent secured; screening and entry into study; baseline data collection (FMPS), randomization into one of the four treatment arms as per the randomization protocol;

- ii. Treatment (T0): all patients will receive a full-mouth professional oral hygiene. Procedures will be performed in the following chronological sequence:
  - A. Place Optragate
  - B. Start the timer for the executive time
  - C. According to the randomization list, patients assigned to the **GBT+** will do professional oral hygiene guided by disclosing plaque (GBT):
- Placement the disclosing plaque agent (Biofilm Discloser® (EMS Electrical Medical Systems SA, CH 1260-Nyon, Switzerland)) on the teeth and rinse with only water;
- Tissue decontamination with Air-flow (Air-flow® Prophylaxis Master EMS, Nyon Switzerland) and erythritol powder (PLUS powder® EMS, Nyon Switzerland);
- Supragingival removal biofilm with Air-flow (Air-flow® Prophylaxis Master EMS, Nyon Switzerland) and erythritol powder (PLUS powder® EMS, Nyon Switzerland);
- Subgingival removal biofilm with Air-flow (Air-flow® Prophylaxis Master EMS, Nyon Switzerland) and erythritol powder (PLUS powder® EMS, Nyon Switzerland);
- Calculus removal with piezoceramic device (Air-flow® Prophylaxis Master EMS, Nyon Switzerland), with a slim tip (PS® EMS, Nyon Switzerland);
- The treatment ends, when all the disclosing plaque has been removed;
- Stop the timer and note the executive time:
- Questionnaire patient and operator;
- Placement of the disclosing plaque agent (Biofilm Discloser® (EMS Electrical Medical Systems SA, CH 1260-Nyon, Switzerland)) on the teeth and rinse with only water;
- Note the FMPS;
- Collection of the pictures.
  - D. According to the randomization list, patients assigned to the **GBT-** will receive professional oral hygiene without the guide by disclosing plaque. The treatment as same as group A without the use of disclosing plaque at the beginning.
  - E. According to the randomization list, patients assigned to the **US+C+** will do traditional professional oral hygiene guided by disclosing plaque:
- Placement the disclosing plaque agent (Biofilm Discloser<sup>®</sup> (EMS Electrical Medical Systems SA,
   CH 1260-Nyon, Switzerland)) on the teeth and rinse with only water;
- Calculus removal with piezoceramic device (Air-flow® Prophylaxis Master EMS, Nyon Switzerland), with a slim tip (PS® EMS, Nyon Switzerland);
- Supragingival and subgingival removal biofilm with rubber cup and polish;

- The treatment ends, when all the disclosing plaque has been removed;
- Stop the timer and note the executive time;
- Questionnaire for the patient and the operator;
- Placement of the disclosing plaque agent (Biofilm Discloser® (EMS Electrical Medical Systems SA, CH 1260-Nyon, Switzerland)) on the teeth and rinse with only water;
- Note the FMPS:
- Collection of the pictures.
  - F. According to the randomization list, patients assigned to the **US+C-** will receive professional oral hygiene without the guide by disclosing plaque. The treatment as same as group C without the use of disclosing plaque at the beginning.
  - G. All treatments are made by the same clinician.
  - H. Data collection (FMPS): A PCP-UNC 15 periodontal probe is used on six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) with a gentle probing force by the same clinician. Measurements are rounded to the nearest millimeter.
  - I. Clinical assessment data will be recorded via hard copy CRFs. CRFs will be submitted to a data entry staff member for entry into the statistical database. At the conclusion of the study, such statistical database will be submitted to the statistician for the preparation of the statistical analysis and the final study report.

#### 2. TREATMENTS

Plus Powder and Biofilm Discloser<sup>®</sup> by EMS Electrical Medical Systems SA, CH 1260-Nyon, Switzerland will be delivered to the study center prior study start.

#### **Concomitant Therapy**

A necessary concomitant medication or therapy is permitted as long as it is not excluded in the exclusion criteria. Every medication has to be reported in the CRF (Appendix 1) and in the Concomitant Medication form (Appendix 2). All changes during the study are to be reported in the CRF. Usage of prohibited therapy will lead to the exclusion of the subject.

# **Blinding and Randomization**

Blinding: The statistician will be blinded to the 4 groups identification, and defined as all the possible combination of A-b (treatment) and B-b (DPA usage).

Randomization and allocation concealment: The randomization will be done based on a computer-generated table, using a random blocks randomization algorithm, that links each patient to one of the four treatment combinations

Implementation: The Principal Investigator will be informed immediately of Serious Adverse Events (SAEs), regardless of the causality relationship between the administration of the investigational treatment and the SAE.

# 3. **PROCEDURE**

# Screening and Selection of Subjects

Patients visiting the Department of Dentistry at Brescia University will be asked to participate in this study. Subjects will report to the clinical facility and be screened by the dental examiner to identify those subjects who meet the inclusion/exclusion characteristics. The findings of this initial screening procedure will be recorded on the CRF. Subjects who meet the inclusion/exclusion characteristics and sign an Informed Consent Form will be entered into the study.

# Baseline Oral Soft and Hard Tissue Assessment

All subjects will receive an evaluation of their oral soft and hard tissues. This examination will include an evaluation of the soft and hard palate, gingival mucosa, buccal mucosa, mucogingival fold areas, tongue, sublingual and submandibular areas and the tonsillar and pharyngeal areas. The results of this evaluation will be recorded on the CRF.

#### Clinical Periodontal Evaluation

All patients receiving treatment will be evaluated by the dental examiner for the following assessments

• Full Mouth Plaque Score (FMPS).

All parameters will be recorded in the CRF.

#### Treatment

Patients who have been identified for treatment will be randomized according to a randomization table generated. The entire mouth will be treated (supra/subgingival) in a single session. If the patient has been identified to receive the control treatment, all teeth

present will not receive the application of disclosing agent and will receive directly full-mouth supragingival and intra sulcular biofilm removal with Airflow or rubber cup and full mouth calculus removal. If the patient has been identified to receive the test treatment, he/she will start full mouth with the application of disclosing plaque.

A questionnaire and OHI are administered

#### 4. STATISTICAL ANALYSIS

Data will be described using standard summary statistics such as mean and standard deviations for quantitative variables, absolute counts and proportions for categorical variables. The primary outcome is Residual Plaque Area (RPA). RPA, expressed as proportion (0-1) will be modelled using a beta-regression model.

Results will be expressed as estimates and relative 95% confidence intervals. A significant level of 5% will be used for all the comparisons and all analysis will be performed using R (version 4.2.1 or higher).

#### Sample size determination

Sample size was estimated via Monte Carlo simulation (B=1000 runs). We assumed a beta-regression model for RPA with technique (USB,GBT) and DPA (No,Yes) as man factors, and their interaction. The parameter of interest is the interaction, i.e. if applying the DPA is giving better results depending on the main technique used. Using data from a previous study on RPA we estimated the phi parameter for a beta distribution (phi=55) and assumed a baseline RPA (no DPA in either techniques) of 10%, with a reduction to 2.9% and 1.5% respectively for USB+C+ and GBT+.

Through simulation we evaluated the sample size needed to achieve a power of at least 80% for the test on interaction term assuming a 5% significance level. A sample size of 30 patients in each of the four group (N=120 overall) achieved a 83% power.

#### **Evaluation of Safety**

The following safety variables will be used for the evaluation of safety:

- Adverse events (AE);
- Adverse reactions (AR).

The total number of AEs and the total number of AEs at least possibly related to the study treatment, as well as the total number of patients affected by at least one adverse event will be calculated per treatment group.

The type of AE classified by organ system (according to MedDRA terminology) will be tabulated. Serious and/or unanticipated adverse events and AEs resulting in discontinuation or reduction/withdrawal of the study treatment will be presented separately.

#### Safety analysis set

Safety summaries will be based on the safety analysis set which will consist of all patients who received the test/control treatment.

#### 5. **MONITORING AND AUDIT**

### **Study Monitoring**

The study will be monitored by the Principal Investigator at periodic intervals during the course of the study to ensure that the study is being conducted according to Good Clinical Practice.

The Investigators will be contacted by the PI on a regular basis. On this occasion, the progress of the study will be discussed with the Investigator and the CRFs will be checked for completeness and consistency and to verify compliance with the study protocol.

#### 6. SUBJECT TERMINATION/WITHDRAWAL PROCEDURES

All efforts will be made to determine the reason(s) why a patient is withdrawn from the study. Subjects could be withdrawn from the study if any of the following occur:

- 1. Subject fails to substantially comply with the protocol requirements;
- 2. Subject develops a serious adverse reaction. The Study Investigator will immediately notify the PI and information will be recorded on a Serious Adverse Event Form (Appendix 3);
- 3. Subject elects to terminate participation in the study. Participation in the study is voluntary. A subject has the right to withdraw from the study at any time for any reason.

The Investigator may terminate the study at any time if the risk-benefit ratio is no longer favourable. Before discontinuation, the Investigator should inform the PI and ask for advice. If the Investigator is concerned about continuation of the study, his/her concerns should be transmitted immediately to the PI.

7. DOCUMENTATION AND DATA MANAGEMENT

Data collection in the case report form (CRF)

All study data will be recorded in the case report forms identified by the subject number. Only the

principal investigator, co-investigators, or designated study personnel may make entries in the

case report forms.

The Investigator has to identify all data that were directly recorded into the CRF and to be

considered to be source data.

The CRFs will be checked for completeness and plausibility by the PI. The Investigator will resolve

any queries.

Investigator Site File (ISF)

The ISF includes all documents that are required for the clinical study. During monitoring, the ISF

will be checked regularly for completeness and actuality. After the clinical trial is finished or stopped,

the ISF has to be stored 15 years in the study center.

**Data Management** 

Data extraction from CRFs into a single, electronic database is performed by examiners.

Discrepancies are to be clarified and corrected by authorized persons by means of documented

data gueries between Statistician and Investigator(s).

After the study is finished and before data are analyzed, a blind data review meeting will be held

between the investigator and the statistician. When the database has been declared to be

complete and accurate, it will be locked. Any changes to the database after this procedure can

only be made by joint written agreement among the clinical trial leader, the trial statistician, and

the co-investigators.

8. ADVERSE EXPERIENCES/EVENTS

Subjects will be informed of any possible adverse reactions which they could experience and will

be instructed to immediately report any event to the investigator. The investigators will record any

and all adverse reactions and report this documentation to the Principal Investigator. In the event

of an adverse experience, emergency or other problems or questions regarding participation in this

study, the subject can contact the following investigators:

for Brescia Site: (Principal Investigator)

Versione 1 del 10/10/2022

12

Adverse Events (AEs) and Serious Adverse Events (SAEs) are defined by the ICH Guideline Medical Device Directive 93/43/EEC and Guidelines on Medical Devices MEDDEVG 2.7/3rev. 3, May 2015 Clinical Investigations: Serious Adverse Event Reporting under Directives 90/385/EEC and 93/42/EEC for Good Clinical Practice (ICH GCP) as follows:

An adverse event (AE) is any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device.

With respect to intensity, adverse events are classified as follows:

- Mild Some awareness of symptoms, but easily tolerated;
- Moderate Symptoms causing enough discomfort to interfere with usual activity;
- Severe Incapacitating event causing inability to work or to perform usual activity.

Adverse events are classified as either non-serious or serious.

# **Serious Adverse Event** (SAE) is an adverse event that:

- a) led to a death;
- b) led to a serious deterioration in health of the subject, that either resulted in:
  - a life-threatening illness or injury, or
  - a permanent impairment of a body structure or a body function, or
  - in-patient hospitalization or prolongation of existing hospitalization, or
  - in medical or surgical intervention to prevent life threatening illness or
  - injury or permanent impairment to a body structure or a body function.
- c) led to fetal distress, fetal death or a congenital abnormality or birth defect.

**Device deficiency:** inadequacy of an investigational medical device related to its identity, quality, durability, reliability, safety or performance. This may include malfunctions, use error, or inadequacy in the information supplied by the manufacturer.

AEs include any clinically significant deterioration of a subject's medical status, after being enrolled and signing an informed consent form. The AE may involve any organs or systems and can be represented by the new onset or the deterioration of a disease, a syndrome, a symptom, a physical

sign, as well as by findings and results of instrumental examinations and laboratory tests. Any medically relevant and untoward change from baseline, including frequency or pattern changes for a fluctuating condition (e.g., migraine), occurring after the administration of investigated treatments is an adverse event. All such occurrences must be recorded and reported accordingly, whether they appear causally related to the study medication, or not.

**Serious Adverse Device Effect** (SADE) is an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

**Unanticipated Serious Adverse Device Effect** (USADE) is a serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report or investigator's brochure (IB).

NOTE: Anticipated SADE (ASADE): an effect which by its nature, incidence, severity or outcome has been previously identified in the risk analysis report or IB.

The following events are considered reportable:

- any SAE;
- any Device Deficiency that might have led to a SAE if:
  - a) suitable action had not been taken or
  - b) intervention had not been made or
  - c) if circumstances had been less fortunate;
- new findings/updates in relation to already reported events.

Reportable events have to be reported by clinical investigators.

#### **Assessment of Causality**

The following criteria are to be used for the assessment of the causal relationship to the test/control treatment. For classification, all criteria of one of the following categories must be met:

#### related, if

- · a timely correlation exists and
- dechallenge and/or rechallenge and
- a biological plausibility exists and
- · other factors are clearly excluded

· a medical report or clinical proof exists;

## possibly related, if

- · a timely correlation exists and
- · dechallenge and/or rechallenge and
- · a biological plausibility exists and
- a medical report or clinical proof does not exist;

# unrelated, if

- · a timely correlation does not exist or is uncertain and
- dechallenge and/or rechallenge does not exist and
- a biological plausibility exists and
- a medical report or a clinical proof does not exist;

#### unknown, if

- not enough information exists for evaluation
- no further contact with reporter possible.

Sound medical/clinical judgment will be applied when assessing the causality and seriousness of the adverse events.

#### **Adverse Event Reporting**

The study center will provide the study participants with emergency telephone numbers for study related support and feedback. The emergency telephone number is operated by either an investigator of the study or by a qualified person designated by the principal investigator. The schedule of reachability of the emergency telephone number will be defined prior to start of the study.

#### Serious Adverse Events

The Investigator shall immediately after awareness (and in any event, not later than within 24 hours after awareness) inform the PI. The Investigator will send the SAE report to the following email address. Appendix 3 has to be used for SAE reporting. Form has to be completed electronically and in English.

# Adverse Events

Adverse events will be assessed by the investigator or designee within 24 hours for severity, relationship to the study product, possible etiologies, and whether the event meets the criteria as a serious adverse event and therefore requires immediate notification to the PI. For data collection purposes, the outcome of all adverse events recorded on the Adverse Reaction section of the CRF will be designated as of the completion of the final evaluation or examination. However, the investigator is responsible for following all adverse events until resolution or until no longer of clinical concern, and providing these data to the PI. At the end of the study, the investigator will report all adverse events (serious and non-serious) to the PI on CRFs. Forms have to be completed electronically and in English.

#### **Pregnancy**

No pregnant women (according to medical history) will intentionally be enrolled in this study. In the event a woman enrolled in this clinical research study becomes pregnant during the course of the study, participation in this study will be terminated upon the clinical staff's notification of the event. The subject's medical records used in this study will be updated to reflect the pregnancy and there will be follow- up contact until the end of the pregnancy to record the outcome in the clinical file.

# 9. ADHERENCE TO PROTOCOL/AMENDMENT(S)

The Investigator will be required to adhere to the final protocol. Any changes to the protocol, except those necessary to eliminate apparent hazards, will require prior approval by the local reviewers through the submission of a protocol amendment. In the event of emergency, the Investigator shall engage any medical procedures that he/she deems appropriate. However, all such procedures must be promptly reported to the PI and Ethical Committee.

The Ethical Committee which granted approval for the study must be notified of all changes in the protocol and must provide written approval if changes are substantial (e.g. increase the risk to the subject, and/or affect the rights of the subject or validity of the investigation, change of/within study population, number of participants or changes of patients' age group).

Departures from eligibility requirements may be allowed on a case-by-case basis by the medical monitor or other authorized sponsor representative. Such departures must be medically and scientifically justified, must be pre-authorized, and must be documented in the CRF and tracked as official eligibility waivers.

#### 10. ADMINISTRATIVE ASPECTS

# **Final Report**

Following the completion of the study, the PI shall prepare a final study report. The final report will include a general description of the conduct of the study including protocol deviations, subject withdrawals, discussion of any adverse events, safety and efficacy data, and statistical analysis of the data. This report will be shared with the Co-investigator at the Participating Centre by the Principal Investigator, and agreed upon parts before being sent to the Sponsor.

#### **Data Retention**

The information in this and any further document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by law or regulations.

In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them.

The files pertaining to this study will be kept by the University-Hospital of Brescia for a period of 15 years from the day of delivery of the final report and will be available for consultation by competent authorities at any time.

The Investigators will retain originals of the approved study protocol, copies of completed CRFs, subjects' participation agreements, relevant source documents and all other supporting documentation related to the study for a period of 5 years. These files must be made available for inspection upon reasonable request by an authorized representative of EMS or the competent authorities.

#### 11. ETHICAL ASPECTS AND REGULATIONS

# **Ethical Conduct of the Study**

This study is to be conducted in accordance with the ethical principles of the Declaration of Helsinki and according to local laws and regulations.

#### Independent Ethics Committee (IEC) and Relevant Authorities

Before starting the study, the study protocol will be subject to review by the Ethical Committee of the University-Hospital of Brescia. As required by law, the study will be notified to authorities if applicable. No subject should be admitted to the study before the Ethical Committees issue their written favourable opinion of the study. Periodic status reports must be reported to the ethics committee at least annually as well as notification of the completion of the study. The investigator

must maintain an accurate and complete record of all reports and documents submitted to and received from the ethics committee according to the ISO 14155:2011 Clinical Investigation of Medical devices for human subjects.

# Subject information and Informed consent form

The purpose and description of the study in lay language, possible adverse reactions, risks and benefits of participation and the subject's right to withdraw without prejudice at any time must be explained to each subject. Each subject must read, understand and sign the informed consent form provided before any study-related procedure.

# Subject data protection and Confidentiality

The name of the subject as well as all other personal data will be kept strictly confidential by the Investigator. If due to medical reasons, it is necessary to identify the subject during the study course, this will be done under medical secrecy.

The subject has given his/her consent before the beginning of the study. In case of withdrawal of this consent subject has to leave the study.

All subjects will agree to verify, by letter, that they participated in this study, if called upon to do so.

#### **New Findings**

Subjects will be informed of any significant new findings related to study products or procedures when they become known during the course of this clinical research study. Such information may affect the subject's decision to continue participation in the study.